CLINICAL TRIAL: NCT01049737
Title: Cardiovascular Risk Factors in Patients With Diabetes -a Prospective Study in Primary Care
Acronym: CARDIPP
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Carl Johan Ostgren, Professor, MD PhD, Linkoeping University
Other Study IDs: CARDIPP
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus Type 2; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were drawn in the fasting state and analysed for levels of HbA1c, hs-CRP, cytokines, lipid and lipoprotein status etc. RNA is extracted from whole blood and the PPAR-gamma isoform was determined after RT-PCR and analysis of DNA sequence. Several small vials of plasma and serum are stored for later analysis of different hormones, cytokines and antibodies (when the economy of the project allows this, high priority is antibodies against GAD and islet beta-cells and levels of hormones such as resistin, adiponectin, leptin and markers of inflammation in terms of cytokines as IL-1, IL-6, IL-10). Other genetic polymorphisms of importance for risk assessment will also be analysed when the economy allows this.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to prospectively explore the impact from the different cardiovascular risk factors on early cardiovascular organ damage in 761 middle aged patients with type 2 diabetes.

DETAILED DESCRIPTION:
CARDIPP (Cardiovascular Risk factors in Patients with Diabetes - a Prospective study in Primary care) was launched in 2005 with the aim of identifying markers for cardiovascular disease to facilitate earlier and individually adjusted intervention in middle aged patients with type 2 diabetes. The patients in CARDIPP were consecutively recruited from primary health care centres in the counties of Östergötland and Jönköping, Sweden from November 2005 through December 2008. The study enrolled 761 patients with type 2 diabetes, aged 55-65 years and the participation in the study was performed as an extended annual follow up. Blood pressure was measured as the average of three seated measurements taken 1 minute apart and standard anthropometric and clinic evaluations were performed including measurement of waist circumference and sagittal abdominal diameter which is a new and promising measurement of abdominal obesity that may serve as a surrogate marker of insulin sensitivity. We also obtained a recording of 24-hour ambulatory blood pressure. The patients filled out a detailed questionnaire for evaluation of life style factors and exercise habits. Pedometer-determined ambulatory activity for three consecutive days in combination with the questionnaires was used for quantification of daily physical activity.

The cardiovascular investigations were performed at the Department of Physiology, Linköping University Hospital and at County Hospital Ryhov, Jönköping, Sweden. The patients were subjected to cardiac ultrasonography for calculation of left ventricular mass and ejection fraction as well as diastolic cardiac function. Measurement of the carotid, femoral and radial pulse pressure wave form is performed by aid of tonometry, with pressure wave analysis and calculation of central blood pressure. Furthermore, pulse wave velocity in both central elastic and muscular peripheral arteries is defined as an index of arterial wall stiffness. The intima-media thickness (IMT) and the lumen diameter (LD) of the carotid arteries were evaluated using a B-mode ultrasound.

CARDIPP-R comprises a re-investigation of the cohort four years after the completion of the baseline examination and will thus start in November 2009 and will be completed by 2012. In CARDIPP-R, all participants from the baseline study will be invited to the re-investigation. The CARDIPP-R study protocol for the cardiac ultrasonography, the carotid ultrasonographic investigations and tonometry for measurements of the carotid, femoral and radial pulse pressure wave form and pulse wave velocity will follow the CARDIPP baseline protocol.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes

Exclusion Criteria:

* Not able to understand Swedish

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients in CARDIPP were consecutively recruited from primary health care centres in the counties of Östergötland and Jönköping, Sweden from November 2005 through December 2008. The study enrolled 761 patients with type 2 diabetes, aged 55-65 years and the participation in the study was performed as an extended annual follow up.
Sampling Method: Non-Probability Sample
Enrollment: 761 (Actual)
Dates: Start 2005-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass index by cardiac ultrasonography, Intima media thickness by carotid ultrasonographic investigation and tonometry for measurements of the carotid, femoral and radial pulse pressure wave form and pulse wave velocity | 4 years after baseline investigation

SECONDARY OUTCOMES:
Cardiovascular morbidity and mortality | 8-12 years after baseline investigation

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Östgren, PhD, Study Director — Linkoeping University; Fredrik H Nyström, Professor, Principal Investigator — Linkoeping University; Toste Länne, Professor, Principal Investigator — Linkoeping University; Jan Engvall, PhD, Principal Investigator — Linkoeping University; Torbjörn Lindström, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Department of Medical and Health Sciences, Linköping University, Linköping, Sweden

REFERENCES:
- [Result] Dahlen EM, Lanne T, Engvall J, Lindstrom T, Grodzinsky E, Nystrom FH, Ostgren CJ. Carotid intima-media thickness and apolipoprotein B/apolipoprotein A-I ratio in middle-aged patients with Type 2 diabetes. Diabet Med. 2009 Apr;26(4):384-90. doi: 10.1111/j.1464-5491.2009.02693.x. PMID 19388968
- [Result] Wijkman M, Lanne T, Engvall J, Lindstrom T, Ostgren CJ, Nystrom FH. Masked nocturnal hypertension--a novel marker of risk in type 2 diabetes. Diabetologia. 2009 Jul;52(7):1258-64. doi: 10.1007/s00125-009-1369-9. Epub 2009 Apr 25. PMID 19396423
- [Derived] Davidson LT, Chisalita SI, Gauffin E, Engvall J, Ostgren CJ, Nystrom FH. Plasma copeptin independently predicts cardiovascular events but not all-cause mortality in patients with type 2 diabetes: a prospective observational study. Nutr Metab Cardiovasc Dis. 2025 Nov;35(11):104158. doi: 10.1016/j.numecd.2025.104158. Epub 2025 May 19. PMID 40617713
- [Derived] Vergara M, Ostgren CJ, Nystrom FH, Israelsson H. Sense of vitality is associated with cardiovascular events in type 2 diabetes independently of traditional risk factors and arterial stiffness. Diabet Med. 2023 Feb;40(2):e14938. doi: 10.1111/dme.14938. Epub 2022 Aug 30. PMID 36039920
- [Derived] Johansson MA, Vavruch C, Ostgren CJ, Nystrom FH. Circulating TNFrII levels predict incidence of ischemic heart disease and total mortality, independently of intima media thickness and pulse wave velocity in male with type 2 diabetes. Heart Vessels. 2021 Oct;36(10):1591-1596. doi: 10.1007/s00380-021-01857-4. Epub 2021 Apr 19. PMID 33871700
- [Derived] Vavruch C, Nowak C, Feldreich T, Ostgren CJ, Sundstrom J, Soderberg S, Lind L, Nystrom F, Arnlov J. Using proximity extension proteomics assay to discover novel biomarkers associated with circulating leptin levels in patients with type 2 diabetes. Sci Rep. 2020 Aug 4;10(1):13097. doi: 10.1038/s41598-020-69473-2. PMID 32753620
- [Derived] Chisalita SI, Wijkman M, Davidson LT, Spangeus A, Nystrom F, Ostgren CJ. Toe brachial index predicts major acute cardiovascular events in patients with type 2 diabetes independently of arterial stiffness. Diabetes Res Clin Pract. 2020 Mar;161:108040. doi: 10.1016/j.diabres.2020.108040. Epub 2020 Jan 29. PMID 32006647
- [Derived] Blomstrand P, Sjoblom P, Nilsson M, Wijkman M, Engvall M, Lanne T, Nystrom FH, Ostgren CJ, Engvall J. Overweight and obesity impair left ventricular systolic function as measured by left ventricular ejection fraction and global longitudinal strain. Cardiovasc Diabetol. 2018 Aug 14;17(1):113. doi: 10.1186/s12933-018-0756-2. PMID 30107798
- [Derived] Radholm K, Tengblad A, Dahlen E, Lanne T, Engvall J, Nystrom FH, Ostgren CJ. The impact of using sagittal abdominal diameter to predict major cardiovascular events in European patients with type 2 diabetes. Nutr Metab Cardiovasc Dis. 2017 May;27(5):418-422. doi: 10.1016/j.numecd.2017.02.001. Epub 2017 Feb 16. PMID 28390663
- [Derived] Wijkman M, Lanne T, Ostgren CJ, Nystrom FH. Aortic pulse wave velocity predicts incident cardiovascular events in patients with type 2 diabetes treated in primary care. J Diabetes Complications. 2016 Sep-Oct;30(7):1223-8. doi: 10.1016/j.jdiacomp.2016.06.008. Epub 2016 Jun 19. PMID 27400814
- [Derived] Jennersjo P, Guldbrand H, Bjorne S, Lanne T, Fredrikson M, Lindstrom T, Wijkman M, Ostgren CJ, Nystrom FH. A prospective observational study of all-cause mortality in relation to serum 25-OH vitamin D3 and parathyroid hormone levels in patients with type 2 diabetes. Diabetol Metab Syndr. 2015 Jun 12;7:53. doi: 10.1186/s13098-015-0049-9. eCollection 2015. PMID 26078787
- [Derived] Vavruch C, Lanne T, Fredrikson M, Lindstrom T, Ostgren CJ, Nystrom FH. Serum leptin levels are independently related to the incidence of ischemic heart disease in a prospective study of patients with type 2 diabetes. Cardiovasc Diabetol. 2015 May 22;14:62. doi: 10.1186/s12933-015-0208-1. PMID 25994184
- [Derived] Dahlen EM, Tengblad A, Lanne T, Clinchy B, Ernerudh J, Nystrom FH, Ostgren CJ. Abdominal obesity and low-grade systemic inflammation as markers of subclinical organ damage in type 2 diabetes. Diabetes Metab. 2014 Feb;40(1):76-81. doi: 10.1016/j.diabet.2013.10.006. Epub 2013 Nov 26. PMID 24290615
- [Derived] Dahlen EM, Bjarnegard N, Lanne T, Nystrom FH, Ostgren CJ. Sagittal abdominal diameter is a more independent measure compared with waist circumference to predict arterial stiffness in subjects with type 2 diabetes--a prospective observational cohort study. Cardiovasc Diabetol. 2013 Mar 28;12:55. doi: 10.1186/1475-2840-12-55. PMID 23536999
- [Derived] Wijkman M, Lanne T, Grodzinsky E, Ostgren CJ, Engvall J, Nystrom FH. Ambulatory systolic blood pressure predicts left ventricular mass in type 2 diabetes, independent of central systolic blood pressure. Blood Press Monit. 2012 Aug;17(4):139-44. doi: 10.1097/MBP.0b013e328355fdfb. PMID 22735793
- [Derived] Jennersjo P, Ludvigsson J, Lanne T, Nystrom FH, Ernerudh J, Ostgren CJ. Pedometer-determined physical activity is linked to low systemic inflammation and low arterial stiffness in Type 2 diabetes. Diabet Med. 2012 Sep;29(9):1119-25. doi: 10.1111/j.1464-5491.2012.03621.x. PMID 22364114
- [Derived] Jennersjo PE, Wijkman M, Wirehn AB, Lanne T, Engvall J, Nystrom FH, Ostgren CJ. Circadian blood pressure variation in patients with type 2 diabetes--relationship to macro- and microvascular subclinical organ damage. Prim Care Diabetes. 2011 Oct;5(3):167-73. doi: 10.1016/j.pcd.2011.04.001. Epub 2011 May 5. PMID 21546328